CLINICAL TRIAL: NCT02958371
Title: Effect of Choice on Food Pleasure Using fMRI
Acronym: PLEASIN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UMR 914 PNCA - AgroParisTech, INRA, Université Paris-Saclay (Unknown); UR370 QuaPA AgroRésonance - INRA Saint-Génès-Champanelle (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHU- 287
Record Dates: First submitted 2016-10-18; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteers
Keywords: Functional magnetic resonance imaging; Taste; Feeding behavior; Choice behavior
MeSH Terms: conditions — Feeding Behavior

ARMS (1):
- fMRI (Experimental): The study consists in a fMRI experiment intended to observe the effect of the presence of choice on brain activity following consumption of a fruit-flavored drink, compared to the brain activity when the same drink is consumed without choice.
  Interventions: Procedure: fMRI; Behavioral: fruit-flavored drink ingestion

INTERVENTIONS:
Procedure: fMRI
Behavioral: fruit-flavored drink ingestion

SUMMARY:
Previous studies have suggested that consumers who can choose what to eat could find food more pleasant, and consume more of that food, than when in absence of choice. However cognitive mechanisms that could explain the effect of choice have not been investigated. The study consists in a fMRI experiment intended to observe the effect of the presence of choice on brain activity following consumption of a fruit-flavored drink, compared to the brain activity when the same drink is consumed without choice. It is suggested that consumers will appreciate drinks they chose better, and that the activity in gustatory and reward regions will change accordingly to changes in declared food pleasure.

DETAILED DESCRIPTION:
The study will include one inclusion session (S1), one out-of-the-magnet tasting session (S2), and one fMRI session (S3). For all sessions, study drinks used are fruit-flavored drinks and fruit juices available on the French market. All subjects will undergo the same protocol, except for the choice of the three study drinks that will be done individually.

S1. After the inclusion/exclusion criteria have been verified, the subjects will perform tests to verify their gustatory/olfactory functions (four basic tastes testing and ETOC test). They will then taste study drinks, blindly, and rate perceived pleasantness.

S2. The out-of-the-magnet tasting session will include three parts:

S2.1 - familiarization with the study procedures. Subjects will be placed in conditions mimicking the fMRI session: they will be asked to lie in supine position, head placed in a false head coil, with the gustometer fixed above their mouth and a video screen visible to them to deliver instructions (visual paradigm created using E-Prime). They also will be given a rolling wheel to collect feedback. The rest of the session will be spent in this position. Subjects will then taste the whole range of study drinks (each drink twice, in a randomized order) and rate their pleasantness on visual analog scales (VAS).

S2.2. - learning picture-drink associations. Three drinks will be chosen based on the ratings given during the first part of the session (three equally appreciated, well-liked (VAS score >50) drinks). Subjects will then taste these three drinks repeatedly while observing abstract pictures. The objective of this sequence is to learn 3 picture-drink pairs.

S2.3 - associative learning verification. Subjects will taste each of the three drinks and choose the picture to which each drink has been associated. If they fail once, the S2.2 and S2.3 sequences will be repeated. If they fail to learn associations at the second verification, they will be excluded form the study.

S3. The fMRI session's objective is to study cognitive correlates of choice. Subjects will be placed in a 3Tesla fMRI scanner, with the gustometer, visual screen and rolling wheel available as in the S2. The functional fMRI scan will be done using high-resolution protocol (1,5*1,5*1,8mm) covering prefrontal, subcortical and occipital brain areas. Subjects will undergo 80 tastings. In 50% of tastings, they will view the three previously learned pictures and freely choose one of them, then receive 1ml of the drink associated with that picture. In the other 50% of tastings, the picture-drink pair will be received without the possibility to choose. The "no choice" tastings will be computed according to the results of "choice" tastings so that each drink will be consumed the same amount of times in "choice" and "no choice" context.

ELIGIBILITY:
Inclusion Criteria:

* - French resident
* French-speaking
* 18-30 years old
* BMI between 18 and 25kg/m2
* stable weight for at least 3 months
* non-smokers
* favorable results at the study questionnaires (TFEQ, gustatory test, ETOC test)

Exclusion Criteria:

* - unwilling to participate in the study
* minors or adults under guardianship/custody
* subjects without social security
* subjects with a cold
* anosmia or ageusia
* disgust for study products
* allergies to study products
* history of neurologic or psychiatric pathologies
* subjects undergoing exclusion period after another study
* subjects with a counter-indication to undergo an fMRI scan
* subjects on medication

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Estimated)
Dates: Start 2016-11; Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
BOLD signal recorded in the orbitofrontal cortex | at 2 weeks of study

SECONDARY OUTCOMES:
Liking scores measured by the Visual analog scales | at 1 week of study
Liking scores measured by the Visual analog scales | at 2 weeks of study
Number of times each drink was chosen by the subjects | at 2 weeks of study
BOLD signal recorded in the gustatory cortex | at 2 weeks of study
BOLD signal recorded in the insula, frontal operculum and the subcortical regions | at 2 weeks of study

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice CLAISE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France